CLINICAL TRIAL: NCT01087944
Title: Tolerability and User Handling Study of an Autoinjector to Administer 180 µg/0.5 mL Peginterferon Alfa-2a (Pegasys, PEG-IFN)
Brief Title: A Study of Administration of Peginterferon Alfa-2a [Pegasys] by Autoinjector Versus Pre-filled Syringe in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP25154
Record Dates: First submitted 2010-03-09; First posted 2010-03-16 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

ARMS (2):
- 1 (Experimental): Peginterferon via auto-injector device.
  All participants will receive Peginterferon in a cross-over design.
  Interventions: Device: Autoinjector
- 2 (Active Comparator): Peginterferon via pre-filled syringe.
  All participants will receive Peginterferon in a cross-over design.
  Interventions: Device: Pre-filled syringe

INTERVENTIONS:
Device: Autoinjector — Participants received Peginterferon alfa-2a 180 microgram subcutaneously once a week by autoinjector for 3 weeks.
  Arms: 1
Device: Pre-filled syringe — Participants received Peginterferon alfa-2a 180 microgram subcutaneously once a week by pre-filled syringe for 3 weeks.
  Arms: 2

SUMMARY:
This randomized, cross-over, open label study will compare the tolerability and handling of application of peginterferon alfa-2a [Pegasys] by autoinjector versus pre-filled syringe in patients with chronic hepatitis C, either on treatment with peginterferon alfa-2a for at least 12 weeks or treatment-naïve for peginterferon alfa-2a. Patients will be randomized to self-injection of 180mcg peginterferon alfa-2a once a week using either an autoinjector or a prefilled syringe for 3 weeks, then switch to use the other method of injection for another 3 weeks. Anticipated time on study treatment is 6 weeks. Target sample size is <100 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* chronic hepatitis C
* on treatment with peginterferon alfa-2a for >/= 12 weeks at baseline, or treatment-naïve for peginterferon alfa-2a

Exclusion Criteria:

* history or evidence of decompensated liver disease
* autoimmune hepatitis
* hypersensitivity to peginterferon alfa-2a or any of its components
* concomitant treatment that requires administration by self-injection, or prior use of an autoinjector

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (12):
  - Los Angeles, California
  - Bradenton, Florida
  - Orlando, Florida
  - Marietta, Georgia
  - Framingham, Massachusetts
  - Newark, New Jersey
  - Vineland, New Jersey
  - New York, New York
  - Poughkeepsie, New York
  - Asheville, North Carolina
  - Columbia, South Carolina
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 participant's data were included from USA (10 centers). The inclusion period was between 11th March 2010 and 28th May 2010.
Pre-assignment Details: This was a two-arm, randomized, crossover study in adult participants with hepatitis C infection. Participants were randomly assigned to one of two groups, in which they received injections by either pre-filled syringe (PFS) or autoinjector (AI) for the first 3 weeks and then switched to the other injection method for an additional 3 weeks.
Groups:
- Sequence 1 (Auto-Injector Then Pre-filled Syringe): Participants received Peginterferon alfa-2a (PEG-IFN) 180 microgram (mcg) /0.5 milliliter (mL) subcutaneously once a week using autoinjector from Week 1-3 in Treatment Period 1 and using pre-filled syringe from Week 4-6 in Treatment Period 2.
- Sequence 2 (Pre-filled Syringe Then Auto-Injector): Participants received PEG-IFN 180 mcg /0.5 mL subcutaneously once a week using pre-filled syringe from Week 1-3 in Treatment Period 1 and using autoinjector from Week 4-6 in Treatment Period 2.
Period: Period 1 (Week 1-3)
Arm/Group | Sequence 1 (Auto-Injector Then Pre-filled Syringe) | Sequence 2 (Pre-filled Syringe Then Auto-Injector)
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2 (Week 4-6)
Arm/Group | Sequence 1 (Auto-Injector Then Pre-filled Syringe) | Sequence 2 (Pre-filled Syringe Then Auto-Injector)
Started | 29 | 30
Completed | 29 | 28
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who received at least one injection.
Groups:
- Overall: Participants received PEG-IFN alfa-2a 180 mcg SC once a week either AI or PFS for the first 3 weeks and then switched to the other method of injection for an additional 3 weeks. Participants also received ribavirin according to standard of care per the investigator's judgment.
Arm/Group | Overall
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Peginterferon Alfa-2a Administration by Autoinjector
Description: The feasibility of PEG-INF administration by AI was assessed by Injection Method Observational Survey questions, based on following pre-defined questions using a "Yes" or "No" response: 1) Did the participant exhibit any nervousness prior to the injection? 2) Did the participant exhibit any difficulty initiating the injection? 3) Did the participant appear confident performing the injection? 4) Did the participant follow the instructions for performing the injection without the need for additional instructions or guidance? 5) Did the participant experience any technical problems with the device or syringe during the injection? 6) Did the participant withdraw the device/syringe before the injection was complete? 7) Did the participant exhibit any visible pain or physical discomfort? 8) Did the participant appear to be satisfied using the device or syringe? 9) Did the participant exhibit any frustration using the syringe or device?
Time Frame: Week 1, Day 1 (Baseline), Week 2 (Day 8 ± 2 days), Week 3 (Day 15 ± 2 days), Week 4 (Day 22 ± 2 days), Week 5 (Day 29 ± 2 days), Week 6 (Day 36 ± 2 days)
Population: The intent-to-treat (ITT) population included all participants who received at least one injection
Measure: Number; unit: participants
Groups:
- Autoinjector: The AI group includes results from Weeks 1-3 for participants in Treatment Group A (Participants received 180 mcg/0.5 mL PEG-IFN subcutaneously once a week by AI for Weeks 1-3, followed by PFS for Weeks 4-6) and results from Weeks 4-6 for participants in Treatment Group B (Participants received 180 mcg/0.5 mL PEG-IFN subcutaneously once a week by PFS for the Weeks 1-3, followed by AI for Weeks 4-6)
- Pre-filled Syringe: The PFS group includes results from Weeks 1-3 for participants in Treatment Group B (Participants received 180 mcg/0.5 mL PEG-IFN subcutaneously once a week by PFS for the Weeks 1-3, followed by AI for Weeks 4-6)and results from Weeks 4-6 for participants in Treatment Group A (Participants received 180 mcg/0.5 mL PEG-IFN subcutaneously once a week by AI for Weeks 1-3, followed by PFS for Weeks 4-6)
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants
  Injection 1, Nervousness, Yes | 11 | 14
  Injection 1, Nervousness, No | 49 | 45
  Injection 2, Nervousness, Yes | 0 | 3
  Injection 2, Nervousness, No | 58 | 56
  Injection 3, Nervousness, Yes | 1 | 2
  Injection 3, Nervousness, No | 56 | 57
  Injection 1, Difficulty initiating, Yes | 7 | 10
  Injection 1, Difficulty initiating, No | 53 | 49
  Injection 2, Difficulty initiating, Yes | 0 | 2
  Injection 2, Difficulty initiating, No | 58 | 57
  Injection 3, Difficulty initiating, Yes | 0 | 2
  Injection 3, Difficulty initiating, No | 57 | 57
  Injection 1, Confidence, Yes | 58 | 46
  Injection 1, Confidence, No | 2 | 13
  Injection 2, Confidence, Yes | 58 | 57
  Injection 2, Confidence, No | 0 | 2
  Injection 3, Confidence, Yes | 57 | 58
  Injection 3, Confidence, No | 0 | 1
  Injection 1, Following instruction, Yes | 58 | 54
  Injection 1, Following instruction, No | 2 | 5
  Injection 2, Following instruction, Yes | 53 | 53
  Injection 2, Following instruction, No | 5 | 6
  Injection 3, Following instruction, Yes | 55 | 56
  Injection 3, Following instruction, No | 2 | 3
  Injection 1, Technical problems, Yes | 7 | 2
  Injection 1, Technical problems, No | 53 | 57
  Injection 2, Technical problems, Yes | 5 | 1
  Injection 2, Technical problems, No | 53 | 58
  Injection 3, Technical problems, Yes | 3 | 3
  Injection 3, Technical problems, No | 54 | 56
  Injection 1, Withdrawal before completion, Yes | 4 | 0
  Injection 1, Withdrawal before completion, No | 56 | 59
  Injection 2, Withdrawal before completion, Yes | 1 | 0
  Injection 2, Withdrawal before completion, No | 57 | 59
  Injection 3, Withdrawal before completion, Yes | 0 | 1
  Injection 3, Withdrawal before completion, No | 57 | 58
  Injection 1, Pain/Discomfort, Yes | 0 | 2
  Injection 1, Pain/Discomfort, No | 60 | 57
  Injection 2, Pain/Discomfort, Yes | 0 | 1
  Injection 2, Pain/Discomfort, No | 58 | 58
  Injection 3, Pain/Discomfort, Yes | 0 | 2
  Injection 3, Pain/Discomfort, No | 57 | 57
  Injection 1, Satisfaction, Yes | 60 | 51
  Injection 1, Satisfaction, No | 0 | 8
  Injection 2, Satisfaction, Yes | 58 | 55
  Injection 2, Satisfaction, No | 0 | 4
  Injection 3, Satisfaction, Yes | 57 | 56
  Injection 3, Satisfaction, No | 0 | 3
  Injection 1, Frustration, Yes | 1 | 2
  Injection 1, Frustration, No | 59 | 57
  Injection 2, Frustration, Yes | 0 | 2
  Injection 2, Frustration, No | 58 | 57
  Injection 3, Frustration, Yes | 0 | 2
  Injection 3, Frustration, No | 57 | 57

2. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Hemoglobin, Albumin and Total Protein
Description: A marked abnormality was defined as a test result which was outside of the marked abnormality range, and which represented a clinically relevant change from baseline of at least the designated amount. The marked reference range for hemoglobin was 110-200 (gram per liter [g/L]), albumin was 30.0-n.d g/L, and total protein was 55-87 g/L. The clinical relevant change (decrease/ increase) for hemoglobin was (15%, 15%), albumin was (20%, n.d) and total protein was (20%, 20%) respectively.
Time Frame: Week 1, Day 1 (Baseline), Week 4 (Day 22 ± 2 days), and Week 6 (Day 36 ± 2 days)
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants
  High Hemoglobin (n=58, 58) | 1 | 0
  Low Hemoglobin (n=58, 58) | 3 | 3
  High Total Protein (n=58, 58) | 0 | 0
  Low Total Protein (n=58, 58) | 0 | 0
  Low Albumin (n=58, 58) | 0 | 0

3. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Hematocrit
Description: A marked abnormality was defined as a test result which was outside of the marked abnormality range, and which represented a clinically relevant change from baseline of at least the designated amount. The marked reference range for hematocrit was 0.31-0.56 fraction. The clinical relevant change (decrease/ increase) for hematocrit was (15%, 15%).
Time Frame: Week 1, Day 1 (Baseline), Week 4 (Day 22 ± 2 days), and Week 6 (Day 36 ± 2 days)
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants
  High Hematocrit (n=58, 58) | 1 | 0
  Low Hematocrit (n=58, 58) | 3 | 1

4. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Platelet, White Blood Cell (WBC), Basophil, Eosinophil, Lymphocyte, Monocyte and Neutrophil
Description: A marked abnormality was defined as a test result which was outside of the marked abnormality range, and which represented a clinically relevant change from baseline of at least the designated amount. The marked reference range for Platelets was 100-550 (10*9/L), for WBC was 3.0-18.0 (10*9/L), for Basophils was 0.00-0.40 (10*9/L), for Eosinophil was 0.00-0.90 (10*9/L), for Lymphocytes was 0.70-7.60 (10*9/L), Monocyte was 0.00-1.70 (10*9/L), and Neutrophil 1.50-9.25 (10*9/L). The clinical relevant change (decrease/increase) for platelet was (30%, 50%), WBC was (30%, 30%), Basophil was (n.d, 100%), Eosinophil was (n.d, 100%), Lymphocyte was (30%, 30%), Monocyte was (n.d, 100%) and Neutrophil was (20%, 20%) respectively.
Time Frame: Week 1, Day 1 (Baseline), Week 4 (Day 22 ± 2 days), and Week 6 (Day 36 ± 2 days)
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants
  High Platelets (n=57, 58) | 0 | 0
  Low Platelets (n=57, 58) | 5 | 3
  High White Blood Cells (n=58, 57) | 0 | 0
  Low White Blood Cells (n=58, 57) | 11 | 9
  High Basophil (n=58, 58) | 0 | 0
  High Eosinophil (n=58, 58) | 0 | 0
  High Lymphocyte (n=58, 58) | 0 | 0
  Low Lymphocyte (n=58, 58) | 5 | 1
  High Monocyte (n=58, 58) | 0 | 0
  High Neutrophil (n=58, 58) | 0 | 0
  Low Neutrophil (n=58, 58) | 20 | 19

5. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Right Blood Cell (RBC)
Description: A marked abnormality was defined as a test result which was outside of the marked abnormality range, and which represented a clinically relevant change from baseline of at least the designated amount. The marked reference range for RBC was 3.80-6.10 (10*12/L). The clinical relevant change (decrease/ increase) for RBC was (15%, 15%).
Time Frame: Week 1, Day 1 (Baseline), Week 4 (Day 22 ± 2 days), and Week 6 (Day 36 ± 2 days)
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants
  High Red Blood Cells (n=57, 57) | 1 | 0
  Low Red Blood Cells (n=57, 57) | 1 | 1

6. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Prothrombin Time (PT) International Normalized Ratio (INR)
Description: A marked abnormality was defined as a test result which was outside of the marked abnormality range, and which represented a clinically relevant change from baseline of at least the designated amount. The marked reference range for PT-INR was n.d.-2.00. The clinical relevant change (decrease/ increase) for PT-INR was (n.d, 30%).
Time Frame: Week 1, Day 1 (Baseline), Week 4 (Day 22 ± 2 days), and Week 6 (Day 36 ± 2 days)
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants | 0 | 0

7. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Serum Glutamic Oxaloacetic Transaminase (SGOT), Serum Glutamic-Pyruvic Transaminase (SGPT), and Alkaline Phosphatase
Description: A marked abnormality was defined as a test result which was outside of the marked abnormality range, and which represented a clinically relevant change from baseline of at least the designated amount. The marked reference range for SGOT was 0-80 (Units Per Litre [U/L]), SGPT was 0-110 U/L, and alkaline phosphatase was 0-220 U/L. The clinical relevant change (decrease/ increase) for SGOT was (n.d, 50%), SGPT was (n.d, 50%), and ALP was (n.d, 50%) respectively.
Time Frame: Week 1, Day 1 (Baseline), Week 4 (Day 22 ± 2 days), and Week 6 (Day 36 ± 2 days)
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants
  High SGOT (n=58, 58) | 4 | 4
  High SGPT (n=58, 58) | 2 | 1
  High Alkaline Phosphatase (n=58, 58) | 0 | 0

8. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Blood Urea Nitrogen (BUN), Chloride, Potassium, Sodium, Calcium, Glucose
Description: A marked abnormality was defined as a test result which was outside of the marked abnormality range, and which represented a clinically relevant change from baseline of at least the designated amount. The marked reference range for BUN was 0.0-14.3 (millimoles per Liter [mmol/L]), Chloride was 95-115 (mmol/L), Potassium was 2.9-5.8 (mmol/L), Sodium was 130-150 (mmol/L), Calcium was 2.00-2.90 (mmol/L), and Glucose was 2.80-11.10 (mmol/L). The clinical relevant change (decrease/ increase) for BUN was (n.d, 50%), Chloride was (7%, 7%), Potassium was (20%, 20%), Sodium was (7%, 7%), Calcium was (10%, 10%), and Glucose was (75%, 75%) respectively.
Time Frame: Week 1, Day 1 (Baseline), Week 4 (Day 22 ± 2 days), and Week 6 (Day 36 ± 2 days)
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants
  High BUN (n=57, 57) | 0 | 0
  High Chloride (n=58, 58) | 0 | 0
  Low Chloride (n=58, 58) | 0 | 0
  High Potassium (n=58, 58) | 0 | 0
  Low Potassium (n=58, 58) | 0 | 0
  High Sodium (n=58, 58) | 0 | 0
  Low Sodium (n=58, 58) | 0 | 0
  High Calcium (n=58, 58) | 0 | 0
  Low Calcium (n=58, 58) | 2 | 2
  High Glucose (n=58, 58) | 0 | 0
  Low Glucose (n=58, 58) | 0 | 0

9. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Creatinine
Description: A marked abnormality was defined as a test result which was outside of the marked abnormality range, and which represented a clinically relevant change from baseline of at least the designated amount. The marked reference range for Creatinine was 0- 154 (micromoles/liter [umol/L]). The clinical relevant change (decrease/ increase) for Creatinine was (n.d, 50%).
Time Frame: Week 1, Day 1 (Baseline), Week 4 (Day 22 ± 2 days), and Week 6 (Day 36 ± 2 days)
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants | 0 | 0

10. Secondary Outcome: Number of Participants With Abnormalities in Pulse Rate, Temperature, and Blood Pressure
Description: The pulse rate, temperature and blood pressure was assessed during a physical examination. Pulse rate was assessed in beats per minute (bpm), temperature was assessed in degree Celsius (°С), and blood pressure was assessed in millimeters of mercury (mmHg). Vital signs were taken while the participant was supine.
Time Frame: as for outcome 1
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants
  High Pulse Rate | 3 | 4
  Low Pulse Rate | 0 | 0
  High Systolic Blood Pressure | 7 | 10
  Low Systolic Blood Pressure | 0 | 0
  High Diastolic Blood Pressure | 9 | 5
  Low Diastolic Blood Pressure | 0 | 0
  High Temperature | 0 | 0
  Low Temperature | 0 | 0

11. Secondary Outcome: Number of Participants With Abnormalities in Electrocardiograms
Description: A 12-lead ECG was recorded after the participant had been in a semi-supine position for at least 10 minutes. Any clinically significant abnormalities noted on an ECG after the first dose of study drug were captured as AEs
Time Frame: Week 1, Day 1 (Baseline), Week 4 (Day 22 ± 2 days), and Week 6 (Day 36 ± 2 days)
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants | 2 | 2

12. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Upto Day 36
Population: The ITT population included all participants who received at least one injection
Measure: Number; unit: participants
Arm/Group | Autoinjector | Pre-filled Syringe
Number analyzed (Participants) | 60 | 59
participants | 34 | 38

ADVERSE EVENTS:
Time Frame: Up to Week 6 (Day 36 ± 2 days)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Autoinjector | Pre-filled Syringe
Serious Adverse Events (participants affected / at risk) | 2/60 | 0/59
Other Adverse Events (participants affected / at risk) | 21/60 | 32/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autoinjector (N=60) | Pre-filled Syringe (N=59)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Autoinjector (N=60) | Pre-filled Syringe (N=59)
Nausea (Gastrointestinal disorders) | 8 | 8
Diarrohea (Gastrointestinal disorders) | 4 | 8
Vomiting (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 8 | 7
Pain (General disorders) | 5 | 5
Pyrexia (General disorders) | 4 | 5
Chills (General disorders) | 3 | 5
Irritability (General disorders) | 3 | 5
Early satiety (General disorders) | 3 | 1
Injection site erythema (General disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Headache (Nervous system disorders) | 4 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.